CLINICAL TRIAL: NCT03036176
Title: "Effects of a Play-based Family Centered Psychomotor/Psychosocial Stimulation on Recovery of Severely Malnourished Children of 6-60 Months of Age During Nutritional Rehabilitation in the Jimma Zone of Ethiopia"
Brief Title: Family Centered Developmental Intervention on Severely Acutely Malnourished Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jimma University (Other); University Ghent (Other); PXL University College (Other)
Responsible Party: Principal Investigator, prof. dr. Marita Granitzer, prof.dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EPFPS-2010
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Severly Acutely Malnourished Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAM intervention group (Other): Children in the intervention group received routine medical treatment and nutritional rehabilitation services in hospital; their primary caregivers were given basic orientations on child care, feeding and nutrition. Children attended play-based stimulation sessions in which trained nurses demonstrated caregivers on how to stimulate the SAM child using play materials and facilities at playroom and playground of the hospital. After discharge from hospital, they were followed up at home and visited three times over a period of six months. During the visits, new play materials were provided and caregivers were shown how to use them to stimulate the SAM child.
  Interventions: Behavioral: Play-based family centered stimulation
- SAM control Group (Other): The control children received routine medical treatment and nutritional rehabilitation services in hospital. Though they had access to playground facilities neither the control children nor their caregivers had access to the playroom materials and the basic orientation on child care, feeding and stimulation.
  Interventions: Other: no intervention

INTERVENTIONS:
Behavioral: Play-based family centered stimulation — Children in the intervention group received routine medical treatment and nutritional rehabilitation services in hospital; their primary caregivers were given basic orientations on child care, feeding and nutrition. Children attended play-based stimulation sessions in which trained nurses demonstrated caregivers on how to stimulate the SAM child using play materials and facilities at playroom and playground of the hospital. After discharge from hospital, they were followed up at home and visited three times over a period of six months. During the visits, new play materials were provided and caregivers were shown how to use them to stimulate the SAM child.
  Arms: SAM intervention group
Other: no intervention — On the other hand, the control SAM group did not receive the guided psychomotor/psychosocial stimulation services although they had access to the playground facilities. Both the intervention and the control groups received all the routine medical care and dietary rehabilitation services at the hospital.
  Arms: SAM control Group

SUMMARY:
Children with severe acute malnutrition (SAM) are at serious risks that compromise their growth and development. Studies have shown the benefits of psychosocial intervention in mitigating the negative consequences of SAM. However, such intervention studies have targeted the critical period in child development and thus focused on children under three years of age. Dietary rehabilitation is usually included as part of the intervention package. Moreover, these young children in such studies customarily obtain more care than older ones and have access to breast milk, more frequent interaction with mother and other caregivers in the family. Therefore, effects of psychosocial interventions targeting such age groups may be different for older children. Much is not known if children older than three years of benefit from similar interventions, and if family-based psychomotor/psychosocial intervention can benefit SAM children in low income contexts such as Ethiopia where access to balanced diet remains hardly possible. In Ethiopia, one of the poorest countries in the world, many children are admitted to hospital for treatment due to SAM. The nutritional rehabilitation unit at hospitals provide dietary treatment to the SAM children who are also treated for related illnesses and complications. Once discharged from hospital, however, the SAM children return to the same poor home environments with inadequate care and unbalanced diets. The main objective of this study was to evaluate the effect of play-based family-centered psychomotor/psychosocial stimulation on linear growth, nutritional status and developmental outcomes of under-six SAM children in the Jimma Zone, south west Ethiopia. This was done by randomly assigning the SAM children admitted to Jimma University's Specialized Referral Teaching Hospital into control and intervention groups. Both groups were receiving the routine medical and dietary treatment services. The intervention group additionally received play-based psychomotor/psychosocial stimulation. Caregivers, supported by periodic visits made to their homes, continued the simulation. Measurements were taken after six months of home follow-up. It was hypothesized that the intervention would significantly improve some of the developmental skills of these children, and that the effect may be age-dependent.

ELIGIBILITY:
SAM children who were admitted for medical treatment and nutritional rehabilitation after being confirmed by physicians to be severely acutely malnourished.

Inclusion criteria were:

1. children between 6 to 60 months of age
2. of Transition Phase i.e., Phase II (no medical complications) and, whose wasting was severe (weight for height or weight for length less than 70% of the median on National Centre for Health Statistics of USA; or
3. with a low mid upper arm circumference (MUAC), i.e., less than 110 mm with a length greater than 65 cm; or,
4. having bilateral pitting edema,

Exclusion criteria were:

SAM children

1. who were completely deaf or blind,
2. who had complications that hinder mobility for play,
3. whose primary caregiver was not able to provide stimulation due to physical or mental disability,
4. who were from far or inaccessible distance for follow-up

Ages: 6 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Language outcome | baseline
  Denver II-Jimma was used to test language outcome & the total number of items successfully performed was counted.
Language outcome | at discharge from the hospital (on average at 2 weeks)
  Denver II-Jimma was used to test language outcome & the total number of items successfully performed was counted.
Language outcome | 6 months after discharge from hospital
  Denver II-Jimma was used to test language outcome & the total number of items successfully performed was counted.
Personal-Social outcome | baseline
  Denver II-Jimma was used to test Personal-social outcome & the total number of items successfully performed was counted.
Personal-Social outcome | at discharge from the hospital (on average at 2 weeks)
  Denver II-Jimma was used to test Personal-social outcome & the total number of items successfully performed was counted.
Personal-Social outcome | 6 months after discharge
  Denver II-Jimma was used to test Personal-social outcome & the total number of items successfully performed was counted.
Fine motor outcome | baseline
  Denver II-Jimma was used to test Fine motor outcome & the total number of items successfully performed was counted.
Fine motor outcome | at discharge from the hospital (on average at 2 weeks)
  Denver II-Jimma was used to test Fine motor outcome & the total number of items successfully performed was counted.
Fine motor outcome | 6 months after discharge
  Denver II-Jimma was used to test Fine motor outcome & the total number of items successfully performed was counted.
Gross motor outcome | baseline
  Denver II-Jimma was used to test Gross motor outcome & the total number of items successfully performed was counted.
Gross motor outcome | at discharge from the hospital (on average at 2 weeks)
  Denver II-Jimma was used to test Gross motor outcome & the total number of items successfully performed was counted.
Gross motor outcome | 6 months after discharge
  Denver II-Jimma was used to test Gross motor outcome & the total number of items successfully performed was counted.
Social-emotional outcome | baseline
  The Ages and Stages questionnaire: Social emotional (ASQ:SE) was used to test Social emotional outcome & a child's total behavior score was obtained by adding up scores on each of the items
Social-emotional outcome | at discharge from the hospital (on average at 2 weeks)
  The Ages and Stages questionnaire: Social emotional (ASQ:SE) was used to test Social emotional outcome & a child's total behavior score was obtained by adding up scores on each of the items
Social-emotional outcome | 6 months after discharge
  The Ages and Stages questionnaire: Social emotional (ASQ:SE) was used to test Social emotional outcome & a child's total behavior score was obtained by adding up scores on each of the items

SECONDARY OUTCOMES:
Linear growth | baseline
  Height/length-for-age z score was used to determine linear growth. For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.
Linear growth | at discharge from the hospital (on average at 2 weeks)
  Height/length-for-age z score was used to determine linear growth. For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.
Linear growth | 6 months after discharge from hospital
  Height/length-for-age z score was used to determine linear growth. For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.
Nutritional status (Weight -for-age) | baseline
  Weight-for-age z score was used to determine nutritional status. A child's weight was measured by using a calibrated electronic weighing scale.
Nutritional status (Weight -for-age) | at discharge from the hospital (on average at 2 weeks)
  Weight-for-age z score was used to determine nutritional status. A child's weight was measured by using a calibrated electronic weighing scale.
Nutritional status (Weight -for-age) | 6 months after discharge from hospital
  Weight-for-age z score was used to determine nutritional status. A child's weight was measured by using a calibrated electronic weighing scale.
Nutritional status (Weight for height/length) | baseline
  Weight-for-height/length z score (for under five children) and body-max-index-for age z score (for children above five years) were used to determine nutritional status.
Nutritional status (Weight for height/length) | at discharge from the hospital (on average at 2 weeks)
  Weight-for-height/length z score (for under five children) and body-max-index-for age z score (for children above five years) were used to determine nutritional status.
Nutritional status (Weight for height/length) | 6 months after discharge from hospital
  Weight-for-height/length z score (for under five children) and body-max-index-for age z score (for children above five years) were used to determine nutritional status.
Nutritional status (Mid-upper-arm circumference) | baseline
  Mid-upper-arm circumference z score was used to determine nutritional status. Mid Upper Arm Circumference (MUAC) was measured with MUAC tape.
Nutritional status (Mid-upper-arm circumference) | at discharge from the hospital (on average at 2 weeks)
  Mid-upper-arm circumference z score was used to determine nutritional status. Mid Upper Arm Circumference (MUAC) was measured with MUAC tape.
Nutritional status (Mid-upper-arm circumference) | 6 months after discharge from hospital
  Mid-upper-arm circumference z score was used to determine nutritional status. Mid Upper Arm Circumference (MUAC) was measured with MUAC tape.

CONTACTS AND LOCATIONS:
Overall Officials: Marita Granitzer, prof. dr., Principal Investigator — Hasselt Univerity

REFERENCES:
- [Derived] Abessa TG, Worku BN, Wondafrash M, Girma T, Valy J, Lemmens J, Bruckers L, Kolsteren P, Granitzer M. Effect of play-based family-centered psychomotor/psychosocial stimulation on the development of severely acutely malnourished children under six in a low-income setting: a randomized controlled trial. BMC Pediatr. 2019 Sep 14;19(1):336. doi: 10.1186/s12887-019-1696-z. PMID 31521161